CLINICAL TRIAL: NCT04351828
Title: The Investigation of Nutritional Status, Intestinal Permeability and Quality of Life in People With Celiac Disease
Brief Title: Intestinal Permeability, Nutritional Status and Quality of Life in Celiac Disease
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Yeşim Öztekin, Principal Investigator, Marmara University
Other Study IDs: 09.2018.359; SAG-C-YLP-121218-0630 (Other Grant/Funding Number: Marmara University, Scientific Research Committee (MU-BAPKO))
Record Dates: First submitted 2020-04-12; First posted 2020-04-17 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Celiac Disease; Nutritional Deficiency; Quality of Life
Keywords: celiac disease; gluten; zonulin; nutritional status; quality of life
MeSH Terms: conditions — Celiac Disease; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5 ml peripheral whole venous blood sample after 8-12 hour fasting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac patients compliant to gluten-free diet (GFD): People with celiac disease who compliant to gluten-free diet (GFD) when they accepted in the study
  Interventions: Procedure: Blood draw once a time
- Celiac patients non-compliant to gluten-free diet(NGFD): People with celiac disease who noncompliant to the gluten-free diet (NGFD) group when they accepted in the study
  Interventions: Procedure: Blood draw once a time

INTERVENTIONS:
Procedure: Blood draw once a time — Investigation of intestinal permeability by measuring serum zonulin levels in blood sample

SUMMARY:
Celiac disease is defined as an autoimmune enteropathy with malabsorption of gluten protein. In recent studies, it has been stated that in individuals diagnosed with celiac disease, intestinal epithelial barrier integrity is impaired. Increased zonulin concentration in blood is considered as an indicator of increased intestinal permeability.

Gluten-free diet is the only treatment of celiac disease. Adherence to gluten free diet provides decreasing of intestinal permeability however gluten free diet has different aspects on nutritional status and health related quality of life in people with celiac disease.

The aim of this study is to determine nutritional status, intestinal permeability and quality of life in people with celiac disease. In the study,it primarily hypothesized that celiac patients noncompliant to gluten-free diet may have increased circulating levels of zonulin and increased intestinal permeability compared to celiac patients compliant to gluten-free diet.

DETAILED DESCRIPTION:
Celiac disease is defined as an autoimmune enteropathy that progresses with malabsorption of gluten protein found in wheat, barley, rye and small intestinal mucosal inflammation in individuals with genetic predisposition. Disruption of intestinal barrier integrity play role in the pathogenesis of celiac disease. Zonulin levels increase in the disruption of intestinal permeability in celiac patients.

At the present, the only treatment of celiac disease is life-long gluten-free diet and it requires strict gluten elimination . With compliance to gluten-free diet, thickening of intestinal mucosal layer, decreasing of villi atrophy and decreasing of transcellular infiltration are observed. In other studies, it was stated that adherence to gluten-free diet can repair intestinal permeability and decrease zonulin levels.

While compliance to gluten-free diet is a key point to prevent progression of the disease, nutritional quality of the gluten-free diet affects nutritional status of patients. Moreover,restricted diets in terms of energy or various nutrients affect health-related quality of life. In studies examining all aspects of celiac disease, it has been stated that health-related factors reduce the quality of life in celiac patients.

In conclusion, this study aims to investigate the presence of intestinal permeability with serum zonulin levels in celiac patients, to evaluate nutritional status of patients with anthropometric measurements and food consumption records, and to determine quality of life of patients with validated celiac disease questionnaire. This study in Turkey, is also first study that investigate all these three factors.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-64,
* To be literate,
* To have positive serological anti tissue transglutaminase immunoglobulin A antibodies value,
* To have a small intestinal biopsy proven celiac disease diagnosis at the time of gastrointestinal endoscopy
* To be volunteer by signing the informed consent form.

Exclusion Criteria:

* To have another autoimmune disease such as type 1 diabetes, psoriasis, hashimoto's thyroiditis, rheumatoid arthritis, systemic lupus erythematosus,
* To be in pregnancy or lactation period,
* Taking probiotic/ prebiotics supplements in the last 2 months,
* Taking antibiotics or non-steroidal antiinflammatory drugs in the last 1 week.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with celiac disease
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Serum zonulin levels of people with celiac disease | 1 day
  Zonulin accepted as an indicator of increased intestinal barrier permeability in previous studies . In this research protocol, zonulin kits were used and zonulin levels were analyzed by sandwich enzyme linked immunosorbent assay (ELISA) method in both celiac patients compliant to gluten free diet group and noncompliant to gluten free diet group.

SECONDARY OUTCOMES:
Dietary intake levels of people with celiac disease | 1 day
  Three-day food consumptions of patients were recorded. Food records of each patient were analyzed in "Nutrition Program, Nutrition Information Systems (BEBIS)" program and daily energy and dietary nutrient intake levels of each patient were calculated.
Body weight, fat and muscle mass measurements of people with celiac disease | 1 day
  Body weight (kg), fat mass (kg) and muscle mass (kg) of each patient were measured with a bioelectrical impedance analysis (BIA) based body composition analyzer.
Body height, waist and hip circumference measurements of people with celiac disease | 1 day
  Certain anthropometric measurements of each patient were taken. Height (cm) was measured with a stadiometer. Tape measurements of waist circumference (cm) and hip circumference (cm) were recorded.
Calculation of waist circumference to hip circumference ratio of people with celiac disease | 1 day
  The ratio of waist circumference to hip circumference was calculated by dividing waist circumference measurement value (cm) to hip circumference measurement value (cm).
Quality of life of people with celiac disease | 1 day
  Celiac disease quality of life questionnaire specific to Turkish celiac population was performed. The questionnaire includes twenty eight questions and total point of questionnaire is between 0-196. Total low point indicates low quality of life, high point indicates high quality of life for people with celiac disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Öztekin, Principal Investigator — Marmara University
Locations (1):
- Marmara University Institute of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajamian M, Steer D, Rosella G, Gibson PR. Serum zonulin as a marker of intestinal mucosal barrier function: May not be what it seems. PLoS One. 2019 Jan 14;14(1):e0210728. doi: 10.1371/journal.pone.0210728. eCollection 2019. PMID 30640940
- [Background] Bai JC, Ciacci C. World Gastroenterology Organisation Global Guidelines: Celiac Disease February 2017. J Clin Gastroenterol. 2017 Oct;51(9):755-768. doi: 10.1097/MCG.0000000000000919. No abstract available. PMID 28877080
- [Background] Burger JPW, de Brouwer B, IntHout J, Wahab PJ, Tummers M, Drenth JPH. Systematic review with meta-analysis: Dietary adherence influences normalization of health-related quality of life in coeliac disease. Clin Nutr. 2017 Apr;36(2):399-406. doi: 10.1016/j.clnu.2016.04.021. Epub 2016 Apr 30. PMID 27179800
- [Background] C D, Berry N, Vaiphei K, Dhaka N, Sinha SK, Kochhar R. Quality of life in celiac disease and the effect of gluten-free diet. JGH Open. 2018 Jun 6;2(4):124-128. doi: 10.1002/jgh3.12056. eCollection 2018 Aug. PMID 30483576
- [Background] Fasano A. Intestinal zonulin: open sesame! Gut. 2001 Aug;49(2):159-62. doi: 10.1136/gut.49.2.159. No abstract available. PMID 11454785
- [Background] Fasano A. Intestinal permeability and its regulation by zonulin: diagnostic and therapeutic implications. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1096-100. doi: 10.1016/j.cgh.2012.08.012. Epub 2012 Aug 16. PMID 22902773
- [Background] Ludvigsson JF, Leffler DA, Bai JC, Biagi F, Fasano A, Green PH, Hadjivassiliou M, Kaukinen K, Kelly CP, Leonard JN, Lundin KE, Murray JA, Sanders DS, Walker MM, Zingone F, Ciacci C. The Oslo definitions for coeliac disease and related terms. Gut. 2013 Jan;62(1):43-52. doi: 10.1136/gutjnl-2011-301346. Epub 2012 Feb 16. PMID 22345659
- [Background] Schumann M, Siegmund B, Schulzke JD, Fromm M. Celiac Disease: Role of the Epithelial Barrier. Cell Mol Gastroenterol Hepatol. 2017 Jan 14;3(2):150-162. doi: 10.1016/j.jcmgh.2016.12.006. eCollection 2017 Mar. PMID 28275682
- [Background] Theethira TG, Dennis M, Leffler DA. Nutritional consequences of celiac disease and the gluten-free diet. Expert Rev Gastroenterol Hepatol. 2014 Feb;8(2):123-9. doi: 10.1586/17474124.2014.876360. PMID 24417260
- [Background] Vici G, Belli L, Biondi M, Polzonetti V. Gluten free diet and nutrient deficiencies: A review. Clin Nutr. 2016 Dec;35(6):1236-1241. doi: 10.1016/j.clnu.2016.05.002. Epub 2016 May 7. PMID 27211234
- [Result] Duerksen DR, Wilhelm-Boyles C, Veitch R, Kryszak D, Parry DM. A comparison of antibody testing, permeability testing, and zonulin levels with small-bowel biopsy in celiac disease patients on a gluten-free diet. Dig Dis Sci. 2010 Apr;55(4):1026-31. doi: 10.1007/s10620-009-0813-5. Epub 2009 Apr 28. PMID 19399613
- [Result] Aksan A, Mercanligil SM, Hauser W, Karaismailoglu E. Validation of the Turkish version of the Celiac Disease Questionnaire (CDQ). Health Qual Life Outcomes. 2015 Jun 19;13:82. doi: 10.1186/s12955-015-0272-y. PMID 26088079
- [Result] Barone M, Della Valle N, Rosania R, Facciorusso A, Trotta A, Cantatore FP, Falco S, Pignatiello S, Viggiani MT, Amoruso A, De Filippis R, Di Leo A, Francavilla R. A comparison of the nutritional status between adult celiac patients on a long-term, strictly gluten-free diet and healthy subjects. Eur J Clin Nutr. 2016 Jan;70(1):23-7. doi: 10.1038/ejcn.2015.114. Epub 2015 Jul 15. PMID 26173865
- [Result] Duerksen DR, Wilhelm-Boyles C, Parry DM. Intestinal permeability in long-term follow-up of patients with celiac disease on a gluten-free diet. Dig Dis Sci. 2005 Apr;50(4):785-90. doi: 10.1007/s10620-005-2574-0. PMID 15844719
- [Result] Fasano A, Not T, Wang W, Uzzau S, Berti I, Tommasini A, Goldblum SE. Zonulin, a newly discovered modulator of intestinal permeability, and its expression in coeliac disease. Lancet. 2000 Apr 29;355(9214):1518-9. doi: 10.1016/S0140-6736(00)02169-3. PMID 10801176
- [Result] Fasano A. Physiological, pathological, and therapeutic implications of zonulin-mediated intestinal barrier modulation: living life on the edge of the wall. Am J Pathol. 2008 Nov;173(5):1243-52. doi: 10.2353/ajpath.2008.080192. Epub 2008 Oct 2. PMID 18832585
- [Result] Hauser W, Gold J, Stallmach A, Caspary WF, Stein J. Development and validation of the Celiac Disease Questionnaire (CDQ), a disease-specific health-related quality of life measure for adult patients with celiac disease. J Clin Gastroenterol. 2007 Feb;41(2):157-66. doi: 10.1097/01.mcg.0000225516.05666.4e. PMID 17245214
- [Result] Hall NJ, Rubin G, Charnock A. Systematic review: adherence to a gluten-free diet in adult patients with coeliac disease. Aliment Pharmacol Ther. 2009 Aug 15;30(4):315-30. doi: 10.1111/j.1365-2036.2009.04053.x. Epub 2009 May 26. PMID 19485977
- [Result] Kabbani TA, Goldberg A, Kelly CP, Pallav K, Tariq S, Peer A, Hansen J, Dennis M, Leffler DA. Body mass index and the risk of obesity in coeliac disease treated with the gluten-free diet. Aliment Pharmacol Ther. 2012 Mar;35(6):723-9. doi: 10.1111/j.1365-2036.2012.05001.x. Epub 2012 Feb 8. PMID 22316503
- [Result] Lammers KM, Lu R, Brownley J, Lu B, Gerard C, Thomas K, Rallabhandi P, Shea-Donohue T, Tamiz A, Alkan S, Netzel-Arnett S, Antalis T, Vogel SN, Fasano A. Gliadin induces an increase in intestinal permeability and zonulin release by binding to the chemokine receptor CXCR3. Gastroenterology. 2008 Jul;135(1):194-204.e3. doi: 10.1053/j.gastro.2008.03.023. Epub 2008 Mar 21. PMID 18485912
- [Result] Leffler DA, Edwards George JB, Dennis M, Cook EF, Schuppan D, Kelly CP. A prospective comparative study of five measures of gluten-free diet adherence in adults with coeliac disease. Aliment Pharmacol Ther. 2007 Nov 1;26(9):1227-35. doi: 10.1111/j.1365-2036.2007.03501.x. PMID 17944737
- [Result] Mishra A, Prakash S, Sreenivas V, Das TK, Ahuja V, Gupta SD, Makharia GK. Structural and Functional Changes in the Tight Junctions of Asymptomatic and Serology-negative First-degree Relatives of Patients With Celiac Disease. J Clin Gastroenterol. 2016 Aug;50(7):551-60. doi: 10.1097/MCG.0000000000000436. PMID 26535478
- [Result] Miranda J, Lasa A, Bustamante MA, Churruca I, Simon E. Nutritional differences between a gluten-free diet and a diet containing equivalent products with gluten. Plant Foods Hum Nutr. 2014 Jun;69(2):182-7. doi: 10.1007/s11130-014-0410-4. PMID 24578088
- [Result] Paganizza S, Zanotti R, D'Odorico A, Scapolo P, Canova C. Is Adherence to a Gluten-Free Diet by Adult Patients With Celiac Disease Influenced by Their Knowledge of the Gluten Content of Foods? Gastroenterol Nurs. 2019 Jan/Feb;42(1):55-64. doi: 10.1097/SGA.0000000000000368. PMID 30688709
- [Result] Rondanelli M, Faliva MA, Gasparri C, Peroni G, Naso M, Picciotto G, Riva A, Nichetti M, Infantino V, Alalwan TA, Perna S. Micronutrients Dietary Supplementation Advices for Celiac Patients on Long-Term Gluten-Free Diet with Good Compliance: A Review. Medicina (Kaunas). 2019 Jul 3;55(7):337. doi: 10.3390/medicina55070337. PMID 31277328
- [Result] Serin, Y., & Akbulut, G. Nutritional Status and Health-Related Quality of Life in Adlt Patients With Celiac Disease. CBU International Conference Proceedings 2018; 6: 952-959. https://doi.org/10.12955/cbup.v6.1277
- [Result] Taetzsch A, Das SK, Brown C, Krauss A, Silver RE, Roberts SB. Are Gluten-Free Diets More Nutritious? An Evaluation of Self-Selected and Recommended Gluten-Free and Gluten-Containing Dietary Patterns. Nutrients. 2018 Dec 3;10(12):1881. doi: 10.3390/nu10121881. PMID 30513876
- [Result] Ukkola A, Maki M, Kurppa K, Collin P, Huhtala H, Kekkonen L, Kaukinen K. Changes in body mass index on a gluten-free diet in coeliac disease: a nationwide study. Eur J Intern Med. 2012 Jun;23(4):384-8. doi: 10.1016/j.ejim.2011.12.012. Epub 2012 Jan 28. PMID 22560391
- [Result] Vojdani A, Vojdani E, Kharrazian D. Fluctuation of zonulin levels in blood vs stability of antibodies. World J Gastroenterol. 2017 Aug 21;23(31):5669-5679. doi: 10.3748/wjg.v23.i31.5669. PMID 28883692
- See also: World Health Organization (WHO) classification of BMI — http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthy-lifestyle/body-mass-index-bmi
- See also: Dietary Guidelines for Turkey (TUBER) — http://dosyasb.saglik.gov.tr/eklenti/10915,tuber-turkiye-beslenme-rehberipdf.pdf